CLINICAL TRIAL: NCT07335952
Title: Proximod, a Selective Sphingosine-1-phosphate Receptor 1 Modulator in Patients With Moderate-to-severe Active Rheumatoid Arthritis: a Double-blind, Randomised, Placebo-controlled, Phase 2 Trial.
Acronym: PROXIMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Director of Rheumatology and Immunology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024PHA083
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: proximod; conventional synthetic disease-modifying antirheumatic drugs
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1:1 ratio to administer proximod 5mg daily, proximod 10mg daily or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (No Intervention): Patients will take placebo daily for three month
- proximod 5mg daily (Experimental): Patients will take proximod 5mg daily for three months
  Interventions: Drug: proximod 5mg daily
- proximod 10mg daily (Experimental): Patients will receive proximod 10mg daily
  Interventions: Drug: proximod 10mg daily

INTERVENTIONS:
Drug: proximod 5mg daily — Patients will take proximod 5mg daily
  Arms: proximod 5mg daily
Drug: proximod 10mg daily — Patients will take proximod 10mg daily
  Arms: proximod 10mg daily

SUMMARY:
The goal of this multicenter, randomized, double-blind, placebo-controlled phase 2 clinical trial is to evaluate the efficacy and safety of proximod in active rheumatoid arthritis patients with inadequate response or intolerance to conventional synthetic disease-modifying antirheumatic drugs (csDMARDs). The main questions it aims to answer are:

Evaluate the efficacy of different doses of proximod in active RA patients who have inadequate response or intolerance to conventional synthetic disease-modifying antirheumatic drugs (csDMARDs), and provide a basis for dose selection in the confirmatory phase III clinical study.

Explore the changes of S1P and SPHK before and after treatment of proximod. Participants will take proximod 5mg/10mg daily or placebo for three months and will be followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 years
2. Diagnosed rheumatoid arthritis (RA) according to the 2010 American College of Rheumatology- European League against Rheumatism classification criteria at least 3 months before screening.
3. Have active RA as defined by ≥ 6 swollen joints (based on 66 joint counts) and ≥6 tender joints (based on 68 joint counts) at screening and baseline.
4. High-sensitivity CRP concentrations equal to or exceeding the upper limit of normal value (ULN) or erythrocyte sedimentation rate (ESR) > ULN
5. Have an inadequate response to ≥ 1 csDMARDs, defined by moderate to high disease activity (DAS28 >3.2, CDAI>2.8, SDAI>3.3).

(1) Patients who received MTX treatment for at least 12 weeks before baseline, with no change in MTX dose (10-25 mg/week) for at least 4 weeks before baseline. For those who cannot tolerate a dose of ≥10 mg/week, a dose of ≥7.5 mg/week can be used.

(2) Patients must discontinue all csDMARDs (excluding MTX) and must not use them during the study period. ① Minocycline, penicillamine, sulfasalazine,hydroxychloroquine, chloroquine, azathioprine, gold preparations, cyclophosphamide, tacrolimus, cyclosporine, Tripterygium wilfordii, etc., taken ≥4 weeks before the first administration of the investigational drug. ② For leflunomide used ≥12 weeks before the first administration of the study drug, cholestyramine (8 g, three times daily for 11 days) or activated charcoal (50 g every 6 hours for 24 hours) can be used for drug elimination. Moreover, the elimination drugs should be discontinued at least 2 weeks before the first administration of the study drug. ③ Other medications must be stopped at least 5 drug half - lives or ≥ 4 weeks before the first dose (whichever is longer).

(3) Patients who have used MTX, discontinued MTX for at least 4 weeks. 6. For biological agents, such as: infliximab: Stop the drug for 8 weeks before the first dose; etanercept and tocilizumab: stop the drug for 4 weeks before the first dose; adalimumab, certolizumab, golimumab and abatacept: stop the drug for 10 weeks; rituximab: stop the drug for 6 month before the first dose.

7. Female patients of childbearing potential and male patients must agree to use an effective method of contraception until at least 6 months after the last dose of Proximod.

8. Sign an informed consent for the clinical study, willingness to comply with the study follow-up schedule and other requirements of the study protocol.

Exclusion Criteria:

1. Allergic to any component of proximod. 2. Class IV according to the Classification of Global Functional Status in Rheumatoid Arthritis or wheelchair/bed-bound.

3. Patients who are using one of the following treatment or medicine.

1. An intra-articular or other injectable corticosteroid within 4 weeks prior to Screening
2. Patients receiving daily corticosteroid treatment at a dosage > 10 mg/day or with an unstable dose within four weeks before inclusion.If glucocorticoids have been discontinued, they should be stopped for at least 2 weeks before the first administration of the study drug.
3. Those who are using non-steroidal anti-inflammatory drugs (except paracetamol) and whose dosage has not been stable within 4 weeks before the first administration of the study drug, or those who cannot continue to take the drug at the original stable dosage during the trial. If they have stopped taking the drug, they need to stop taking the drug for at least 2 days or 5 half-lives (whichever is longer) before the first administration of the study drug.
4. Patients who have received treatment with Iguratimod, interferon (such as Roferon, Intron A, Rebetron, etc.), drugs known to have strong immunosuppressive or immunomodulatory effects (including total Glucosides of Paeony, Tripterygium wilfordii Hook.f, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine, 6 - mercaptopurine, etc.), or technetium [99Tc] methylene diphosphonate injection within 4 weeks before the first administration of the study drug.
5. Use of opioids within 4 weeks before the first administration of the study drug.
6. Oral traditional Chinese medicines for the treatment of RA and other inflammatory diseases within 4 weeks before the first administration of the study drug.
7. Subjects who have received integrin Alpha V antibodies or cell depletion therapy within 3 months before the first administration of the study drug or within 5 half - lives (whichever is longer).
8. Received JAK inhibitors and/or S1P agonists within 5 half - lives or within 2 weeks (whichever is longer).
9. Use of medications that interact with the study drug within 4 weeks or within 5 half - lives (whichever is longer).
10. The subject has received live vaccines or live- attenuated vaccines within 4 weeks.
11. Alcohol abuse or drug abuse, or there is a history of alcohol or drug abuse within 6 months before randomization.
12. Patients who have participated in any interventional clinical trials of drugs or medical devices within the past three months.

4. History or evidence of any of the following diseases:

1. Those with any systemic inflammatory diseases/medical history other than RA (except secondary Sjögren's syndrome), including but not limited to inflammatory bowel disease (including Crohn's disease and ulcerative colitis), psoriatic arthritis, vasculitis, gout, systemic lupus erythematosus, axial spondyloarthritis (including ankylosing spondylitis and non-radiographic axial spondyloarthritis), reactive arthritis, scleroderma, polymyositis, dermatomyositis, fibromyalgia (with currently active symptoms), Felty syndrome.
2. A history of lymphoproliferative diseases, or various signs or symptoms that may indicate lymphoproliferative diseases.
3. The subject has a history of any active malignant tumor or malignant tumor within 5 years before the screening visit, except for skin squamous or basal cell carcinoma, carcinoma in situ of the cervix, or ductal carcinoma in situ of the breast that has been treated and considered cured.
4. Those with a history of recurrent herpes zoster (≥2 episodes), disseminated herpes zoster, or disseminated herpes simplex, or those with a history of herpes zoster or herpes simplex within 2 months before randomization, or patients with risk factors are unsuitable for participation..
5. Patients with active tuberculosis indicated by chest X-ray examination and positive results for TB (T-SPOT.TB test or TB-IGRA)
6. Fundus photography and optical coherence tomography show abnormal and clinically significant findings.
7. Hereditary or acquired immunodeficiency diseases, including immunoglobulin deficiency.
8. Severe hematological diseases (e.g., aplastic anemia, myelodysplastic syndromes) or diseases causing hemolysis or red blood cell reduction (e.g., malaria, hemolytic anemia)
9. Mental or neurological diseases, unwillingness/unability to communicate, or inability to understand study requirements/cooperate with the research team
10. Donation of 400 mL or more blood within the past 3 months, or receipt of blood transfusions
11. Active infections (e.g., chronic pyelonephritis, bronchiectasis, osteomyelitis; excluding nail bed fungal infection) deemed unsuitable by the investigator; major infection episodes requiring oral/intravenous anti-infectives within 14 days prior to baseline; or deep infection history (e.g., abscess, osteomyelitis) within 52 weeks before baseline
12. Uncontrolled diseases, such as diabetes, hyperlipidemia, hypertension, kidney diseases, liver diseases, severe cardiovascular and cerebrovascular diseases (such as heart failure [NYHA III or IV], unstable angina, stroke or transient ischemic attack, myocardial infarction, etc.), respiratory diseases, severe chronic gastrointestinal diseases (such as active or recurrent peptic ulcers), or those who have undergone treatments that may affect drug absorption (such as gastrointestinal surgery) and are unsuitable to participate the study.
13. Patients who have undergone major surgery within 4 weeks prior to enrollment; or are expected to undergo major surgery post-enrollment; or have chronic pain affecting study evaluations; or have a history of organ transplantation 5. During screening, there are any abnormal results that meet the following criteria (no medical supportive treatment [e.g., pharmaceutical agents raising white blood cell count, drugs for anemia, liver protective agent, blood transfusion, etc.] is allowed within 2 weeks before screening):

1) Hemoglobin < 90.0 g/L. 2) White blood cell counts < 2.5×10⁹/L. 3) Absolute neutrophil count < 1.5×10⁹/L. 4) Lymphocytopenia (absolute lymphocyte count < 0.750×10⁹/L). 5) Platelet count < 100×10⁹/L. 6) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), total bilirubin (T-BIL) > 2×upper limit of normal (ULN).

7) eGFR of <60 mL/min/1.73 m². 8) Patients positive for HBsAg. Patients who are positive for anti-HBc antibody and HBV-DNA polymerase chain reaction (PCR) above the lower limit of detection; Patients who are positive for Hepatitis C antibody and the hepatitis C RNA PCR above the lower limit of detection; or positive for Treponema pallidum antibody (TP Ab); or positive test for HIV.

6. Female patients who are pregnant or breastfeeding, or those who plan to pregnant or breastfeed during the study period or within 6 months after the last dose.

7. Other factors that may affect the conduct of this study or the evaluation of its results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving American College of Rheumatology (ACR) 20 response at week 12. | Twelve weeks
  The primary efficacy outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University People's Hospital
Locations (20):
- China (20):
  - Chun Li, Beijing, Beijing Municipality
  - Guixiu Shi, Xiamen, Fujian
  - Yi He, Guangzhou, Guangdong
  - Mingwei Deng, Guangzhou, Guangdong
  - Qingwen Wang, Shenzhen, Guangdong
  - Ling Lei, Nanning, Guangxi
  - Jiashun Zeng, Guiyang, Guizhou
  - Mei Tian, Zunyi, Guizhou
  - Xiaofei Shi, Luoyang, Henan
  - Lingli Dong, Wuhan, Hubei
  - Shulin Song, Yichang, Hubei
  - Jian Wu, Suzhou, Jiangsu
  - Senhua Dai, Pingxiang, Jiangxi
  - Yanmei Wu, Panjin, Liaoning
  - Xuebinwang, Binzhou, Shandong
  - Weiqi Min, Heze, Shandong
  - Hua Zhang, Zaozhuang, Shandong
  - Zili Fu, Taiyuan, Shanxi
  - Wubin Long, Chengdu, Sichuan
  - Huaxiang Wu, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The deidentified IPD will be shared to researchers whose proposed use of the data has been approved.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year after publication with no end date